CLINICAL TRIAL: NCT07211334
Title: Comparison of the Effects of Different Exercise Modalities in Frail Elderly People Care Setting
Brief Title: High Intensity Interval Training Versus Moderate Intensity Continuous Training in Frail Elderly
Acronym: EPAF
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: Essaiclinique_EPAF
Record Dates: First submitted 2025-08-25; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Frail Elderly
Keywords: Frailty; Elderly; High Intensity Interval Training; Moderate Intensity Continuous Training; Motivation for Physical Activity; Support for Changing Behavior Regarding Physical Activity
MeSH Terms: conditions — Frailty | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Exercise Training — Adapted High Intensity Interval Training (HIIT), Moderate-Intensity Continuous training (MICT), therapeutic education workshops to help people become independent regarding their program

SUMMARY:
The assessment and systematic integration of physical activity into the care pathway of frail elderly people is essential to prevent loss of independence and improve the quality of life of this population. This project, which is part of routine care, aims to evaluate the practices and, in particular, the effects of different types of physical exercise currently in use at the Health and Sport Center of the Grenoble Alpes University Hospital. It therefore aims to optimize professional practices without changing the standard care provided to patients. Recommendations regarding intensity during cardiorespiratory endurance training sessions (moderate to high, taking into account emotional factors) are broad and vary greatly in their application depending on the facilities that work with older adults. This project aims to compare the exercise methods used on ergocycle at Health and Sport Center of Grenoble Alpes University Hospital: high-intensity interval training (HIIT) vs. moderate-intensity continuous training (MICT) to reverse the functional decline that occurs in frail older adults.

DETAILED DESCRIPTION:
The aging of the population is accelerating worldwide, with a sharp increase in the number of people aged 65 and over. In France, 21% of the population was aged 65 or over in 2022. Individuals in this age group will represent one-third of the French population by 2050. This demographic growth is due to increased longevity combined with a decline in birth rates. However, this increased longevity can be accompanied by significant challenges, including significant functional disabilities and loss of independence. In fact, a significant proportion of this population, namely 15 to 20% of those over 65, is considered frail and at risk of human and material dependence. People of the same age can have very different physiological states. The concept of frailty allows the investigators to consider the heterogeneity of the elderly population and to differentiate between chronological age and "physiological age," which is probably a better indicator of the ability to engage in physical activity (PA).

Frailty in older adults increases the risk of dependence and mortality when exposed to physiological or psychological stress, thus conferring a high risk of adverse health effects. Criteria for frailty include unintentional weight loss (>5kg in the past year), sedentary lifestyle, fatigue, slow walking speed, and lack of strength, reducing functional reserves and the ability to cope with stress. In addition, functional mobility, which is crucial for performing activities of daily living, is often impaired in frail older adults and increases the risk of falls, loss of independence, and institutionalization. According to the French National Authority for Health (HAS), identifying frailty in older people is important in order to use standardized gerontological assessments to identify modifiable factors contributing to frailty and implement targeted, personalized interventions. Physical factors (such as physical inactivity or malnutrition) or psychological factors (such as depression) are causes of frailty that can be identified by healthcare professionals and addressed through preventive or corrective measures. The HAS therefore strongly recommends that exercise prescriptions and measures to combat sedentary lifestyles in frail elderly people be integrated into the care pathway. The aim of prescribing exercise is, on the one hand, to improve the physical condition and mobility of these patients, which are often impaired, and, on the other hand, to combat sedentary lifestyles, which lead to a vicious circle of physical deconditioning. The results of interventional studies including exercise programs indicate benefits both in terms of physical frailty criteria and quality of life in older adults. While the benefits of conventional physical activity programs following health recommendations are undeniable in this population, not all of them appear to be optimal in terms of reversing frailty. Indeed, the recommendations regarding intensity during cardiorespiratory endurance training sessions in particular (moderate to high, considering affects during exercise) are broad and vary greatly in their application depending on the facilities working with older adults, suggesting the need to individualize practices. At the Health and Sports Center of the Grenoble Alpes University Hospital, in accordance with the recommendations, various effective exercise methods are applied and adapted to the needs of the people being treated (level of exercise tolerance, etc.): high-intensity interval training (HIIT) and moderate-intensity continuous training (MICT). According to the literature, HIIT appears to have greater short-term effects on physical fitness, cardiovascular and metabolic morbidity, and body composition in older adults. It is used at the Health and Sport Center at Grenoble Alpes University Hospital, with adaptations for frail elderly people. However, to the knowledge of investigators, the superiority of HIIT over MICT in terms of cardiorespiratory endurance in frail individuals has not been studied. This project therefore aims to identify the exercise modalities that offer optimal and lasting effects on the cardiorespiratory fitness of frail older adults. Thus, the investigators will compare the ergocycle exercise modalities used at the Health and Sport Center of the Grenoble Alpes University Hospital: high-intensity interval training (HIIT) vs. moderate-intensity continuous training (MICT) to reverse the functional decline that occurs in frail elderly people.

While the effects of regular physical activity are widely beneficial to all groups, it requires a long-term commitment. These are the missions of the Health and Sports Centers. This applies to frail elderly people (sedentary by definition) receiving care at Grenoble Alpes University Hospital. Sedentary lifestyles are the gateway to a vicious cycle of physical deconditioning and frailty. To this end, in line with the practices in place at the Health and Sports Center, the investigators support people's motivation through interviews and therapeutic education workshops. These workshops also allow the investigators to assess sleep quality, which can interfere with physical activity and is correlated with frailty. The investigators therefore hypothesize that the support provided by Health and Sport Center incorporating a HIIT exercise program is more effective than support incorporating a MICT exercise program on cardiorespiratory endurance. The primary outcome: will be the comparative evolution over 24 weeks (from W0 to W24) of cardiorespiratory fitness (VO2peak). The secondary outcome will be comparative changes over 24 weeks (at S0, S8, and S24) of body composition, walking ability (distance, walking speed), grip strength, quadriceps strength, Fried's frailty criteria, health-related quality of life in its physical, psychological, and social dimensions, sleep quality, motivation for physical activity (PA) for health purposes. The investigators will include subjects aged 70 or older meeting at least 1 of 5 frailty criteria according to Fried with no acute illness or recent decompensation that could be aggravated by exercise (at the physician's discretion) who do not object to the analysis of their anonymized data, who are affiliated with social security and are able to use an ergocycle safely. Subjects presenting musculoskeletal disorders and severe neurocognitive conditions that make it impossible to safely use the ergocycle or participate in the exercise program will not not be included as well those participating in other interventional studies or who have recently participated in an interventional study that could influence the results of this study. As participants will receive routine care, they will be considered as patients since they will be identified as frail (3 positive criteria out of 5 according to Fried) or pre-frail (1 to 2 positive criteria out of 5 according to Fried) in the geriatric department of Grenoble Alpes Universitary Hospital (CHUGA) (Prof. Gavazzi) and are referred to the EXPLORASUD Sport and Health Center at CHU Sud (Dr. Coudurier, Dr. Doutreleau) for support through physical activity. The research process described below corresponds to the minimum standards implemented at the Health and Sport Center. It will consist in an inclusion visit allowing to check eligibility criteria (identified as frail or pre-frail in the geriatric department of CHUGA, Prof. Gavazzi) and to get their consent to the use of data. Patients will undergo a series of assessments necessary for physical exercise support. These assessments, carried out as part of routine clinical practice at the Health and Sport Center, consist of measuring cardiorespiratory endurance (maximal progressive exercise test), body composition (bioimpedance analysis), walking ability (distance, walking speed), grip strength and quadriceps strength, health-related quality of life, sleep quality/sleepiness, and motivation for physical activity for health purposes. Depending on their preferences and characteristics (particularly exercise intolerance), patients follow either a HIIT or MICT program. Regardless of the program, each patient will participate for six months, with two months of supervised program at the Health and Sport Center of Grenoble Alpes University Hospital (two to three sessions per week), supplemented by advice on how to continue independently, followed by a four-month program that allows for a high degree of independence (remote or in-person supervision, only once a month). The sessions will take place on an ergocycle, which allows for precise control of exercise intensity (power), and a heart rate monitor and effort perception scales will be used to control physiological intensity and exercise acceptability. For the part of the program carried out independently (during the first 2 months or the following 4 months), equipment may be loaned to the patient in accordance with the practices in force at the Health and Sport Center. Patients following HIIT program will perform high-intensity interval training (>85% of VO2peak) for a total of 50 minutes, three times a week, including two to three supervised sessions in person at the Health and Sport Center. Each session will begin with a 10-minute warm-up at a low intensity (between 30 and 40% of VO2peak), after which patients will complete various phases of intense exercise (>85% of VO2peak) for 30 minutes. Each phase of intense exercise will last between 10 seconds and 1 minute, with a passive recovery time between phases lasting between twice and once the exercise time. At the end of each session, patients will cool down for 10 minutes at the same intensity as the warm-up. In addition to this exercise bike session, they will achieve two muscle strengthening and balance sessions recommended for seniors between each session (at the Health and Sport Center and at home). The APA teacher will clearly explain how to perform these exercises. Patients will be provided with a booklet describing a range of "easy to perform" exercises, which will be demonstrated on the day of the supervised sessions. The APA teacher will ensure that patients understand the exercises properly, adjusting the intensity and duration of the exercise when the perceived difficulty exceeds 5/10 on the WHO perceived exertion scale (0-10 in arbitrary units) and the affects become negative on the affect scale (-5 to 5). Patients following MICT program will perform a continuous training session at an intensity of between 40 and 60% of VO2peak for a total duration of 50 minutes, three times a week, including two to three supervised sessions in person at the Health and Sport Center. Each session will begin with a 10-minute warm-up at a low intensity (between 30 and 40% of VO2peak), after which patients will complete the main part of the session at a moderate intensity (40 to 60% of VO2peak). At the end of each session, patients will cool down for 10 minutes at the same intensity as the warm-up. In addition to this exercise bike session, they will achieve two muscle strengthening and balance sessions recommended for seniors between each session (at the Health and Sport Center and at home). The APA teacher will clearly explain how to perform these exercises. Patients will be provided with a booklet describing a range of "easy to perform" exercises, which will be demonstrated on the day of the supervised sessions. The APA teacher will ensure that patients understand the exercises properly, adjusting the intensity and duration of the exercise when the perceived difficulty exceeds 5/10 on the WHO perceived exertion scale (0-10 in arbitrary units) and the affects become negative on the affect scale (-5 to 5). Support for changing physical activity behavior will be performed according to the practices in place at the Health and Sport Center, a motivational interview will be systematically conducted before any physical activity program implementation. In addition, patients will systematically benefit from therapeutic education workshops. The aim of these workshops is to help people become independent in terms of physical activity. This autonomy will be assessed throughout the program (from W0 to W24) using activity sensors belonging to the service (Polar Unite heart rate monitor) to measure energy expenditure and the number of steps taken each day. In parallel with these measures, we will ask patients to record their physical activities in a logbook to compensate for any inability or refusal on the part of patients to use connected devices. After eight weeks of supervised training and 16 weeks of unsupervised training, patients will benefit a follow-up assessment. All initial assessments will be repeated at 8 and 24 weeks, including the assessment of frailty criteria carried out at the CHUGA Geriatric Department (Prof. Gavazzi) before their inclusion in the exercise program of the Health and Sport Center. After eight weeks of training supervised by an Adapted Physical Activity (APA) teacher, participants will continue to exercise independently according to the exercise methods used during the first two months (HIIT or MICT) in order to assess their ability to maintain physical activity in the medium term. In accordance with the practices in place at the Health and Sport Center, a monthly review (by telephone, in person, questionnaires, etc.) will be carried out on the activities completed by patients and any difficulties they might have encountered. If necessary, temporary support can be provided to try to remove barriers to physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 70 or older;
* Patients meeting at least 1 of 5 frailty criteria (Fried criteria; 2001);
* Patient does not object to the analysis of anonymized data;
* Person affiliated with social security;
* Patient's ability to use an ergocycle safely;
* Patients medically stable patients with no acute illness or recent decompensation that could be aggravated by exercise (at the physician's discretion).

Exclusion Criteria:

* Unstable medical conditions that may be aggravated by physical activity (as determined by a physician)
* Musculoskeletal disorders and severe neurocognitive conditions that make it impossible to safely use the ergocycle or participate in the exercise program
* individuals participating in other interventional studies or who have recently participated in an interventional study that could influence the results of this study
* Persons referred to in Articles L1121-5 to L1121-8 of the public health code (corresponds to all protected persons: pregnant women, women in labor, breastfeeding mothers, persons deprived of their liberty by judicial or administrative decision, persons subject to legal protection measures)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged >70 years are receiving routine care. They are identified as frail (3 positive criteria out of 5 according to Fried) or pre-frail (1 to 2 positive criteria out of 5 according to Fried) in the Geriatric Department of Grenoble Alpes Universitary Hospital (CHUGA) (Prof. Gavazzi) and are referred to the EXPLORASUD Sport and Health Center at CHU Sud (Dr. Coudurier, Dr. Doutreleau) for support through physical activity.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory endurance (VO2peak) | At weeks 0, 8 and 24
  in mL/kg/min with an ergospirometer during a maximal progressive test

SECONDARY OUTCOMES:
Fried's frailty criteria | At weeks 0, 8 and 24
  muscle weakness (grip strength in the lowest 20th percentile), reduced gait speed (< 0.8 m/s), self-reported fatigue, low physical activity levels (< 383 kcal/day for men and < 270 kcal/day for women), unintentional weight loss (> 5% body weight over 12 months)
Weight | At Weeks 0, 8 and 24
  Weight scale in kg
Height | At weeks 0, 8 and 24
  in cm with a measuring rod
Body composition | At weeks 0, 8 and 24
  fat mass, fat-free mass, in kg and as percentages of total body weight with bioelectrical impedance analysis using a standardized body composition analyzer (Tanita BC 418 MA; Tanita Corp., Tokyo, Japan)
Health-related quality of life in its physical, psychological, and social dimensions | At weeks 0, 8 and 24
  European Quality of Life 5 Dimensions 5 Level Version : (best score:11111; worse score:33333), Visual Analogic Score for health (best score:100; worse score:0)
Sleep quality and sleepiness | At weeks 0, 8 and 24
  Pittsburgh Sleep Quality Index (best score : 0; worse score : 21) and Epworth Sleepiness Scale (best score : 0; worse score : 24)
Motivation for physical activity for health purposes | At weeks 0, 8 and 24
  EMAPS Questionnaire : (worse score i.e amotivation : -36; best : autodetermined motivation)

IPD SHARING:
Plan to Share IPD: No